CLINICAL TRIAL: NCT03664882
Title: Phase 3, Single-center, Sequential and Parallel-group, Double-blind, Randomized Study Evaluating the Efficacy and Safety of Fexofenadine Hydrochloride 180 mg (Allegra®/Telfast®) Versus Placebo in Subjects Suffering From Seasonal Allergic Rhinitis With Symptoms Aggravated in Presence of Pollutants
Brief Title: Study Evaluating the Efficacy and Safety of Fexofenadine in Subjects Suffering From Seasonal Allergic Rhinitis in Presence of Pollutants
Acronym: FEXPOLSAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPS15332; U1111-1205-1504 (Other: UTN)
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Rhinitis Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fexofenadine (Experimental): Fexofenadine, single administration
  Interventions: Drug: Fexofenadine M016455
- Placebo (Placebo Comparator): Placebo, single administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fexofenadine M016455 — Pharmaceutical form: tablet Route of administration: oral
  Arms: Fexofenadine
Drug: Placebo — Pharmaceutical form: tablet Route of administration: oral
  Arms: Placebo

SUMMARY:
Primary Objectives:

* To demonstrate that the aggravation of seasonal allergic rhinitis symptoms in the presence of pollutants is observed using an Environmental Exposure Unit.
* To evaluate the efficacy of fexofenadine hydrochloride in subjects suffering from seasonal allergic rhinitis symptoms aggravated in the presence of diesel exhaust particulates.

Secondary Objective:

To evaluate the safety of a single dose of fexofenadine hydrochloride 180 mg.

DETAILED DESCRIPTION:
The total study duration per subject is expected to last up to 4.5 months, depending on the timing of the screening visit.

ELIGIBILITY:
Inclusion criteria:

* Males or females between the ages of 18 and 65 suffering from seasonal allergic rhinitis provoked by ragweed pollen.
* Having a 2-year history of seasonal allergic rhinitis with positive skin prick test to ragweed allergen at screening with a wheal diameter at least 3 mm larger than that produced by the negative control.
* Subjects with antecedents of allergic seasonal allergic rhinitis symptom aggravation when exposed to pollen and air pollutants (i.e., cleaning products, diesel, paints).
* Subjects having a total nasal symptom score ≥3 in Period 1 (Visit 2).

Exclusion criteria:

* History of anaphylaxis to ragweed pollen.
* History of asthma. Mild asthmatics treated only with pro re nata short-acting beta2-agonists, 2 doses or less per week can be enrolled.
* History of chronic sinusitis.
* History of systemic disease affecting the immune system.
* Evidence of any active or suspected bacterial, viral, fungal or parasitic infections within 30 days prior to allergen challenge.
* Any history of Grade 4 anaphylaxis due to any cause as defined by the Common Terminology Criteria for Adverse Event grading criteria ("Life threatening consequences: urgent intervention indicated").
* Presence or history of drug hypersensitivity to fexofenadine.
* Subjects receiving build-up injections of pollen allergen immunotherapy (those on stable maintenance dosing can be included).
* Subjects taking any forbidden treatments/nutriments.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | From hour 0 to hour 12 in Period 1 and Period 2
  Assessed by measuring change in the area under the curve (AUC) of the TNSS during Period 1 and 2
TNSS | From hour 2 to hour 12 in Period 3
  Assessed by measuring change in the AUC of the TNSS from hour 2 (planned time of investigational medicinal product administration) to hour 12 in Period 3

SECONDARY OUTCOMES:
Total symptom score (TSS) | From hour 2 to hour 12 in Period 3
  Assessed by measuring change in the AUC of TSS from hour 2 (planned time of investigational medicinal product administration) to hour 12
Individual symptom score | From hour 2 to hour 12 in Period 3
  Assessed by measuring the change in AUC of individual symptom score from hour 2 (planned time of investigational medicinal product administration) to hour 12
TNSS | From hour 2 to hour 12 in Period 3
  Assessed by change in TNSS by time point from hour 2 to hour 12
Adverse events | Up to 4.5 months
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number, Canada, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org